CLINICAL TRIAL: NCT04669652
Title: Will Piezo-ICSI Increase Fertilization Rates Compared to Conventional ICSI? A Prospective Randomized Sibling Study.
Brief Title: Evaluating Piezo-ICSI. - The EPI Study.
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Study on hold
Sponsor: Vitrolife (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4026 - EPI
Record Dates: First submitted 2020-12-01; First posted 2020-12-17 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: IVF; Infertility
Keywords: ICSI; Fertilization; Piezo-ICSI; Oocyte; Blastocyst rate
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: A sibling study randomizing oocytes to 2 study groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICSI (No Intervention): Traditional microinjection (ICSI) is performed on oocytes.
- Piezo-ICSI (Experimental): Microinjection (ICSI) is performed using the Piezo-ICSI technique.
  Interventions: Device: Piezo-ICSI

INTERVENTIONS:
Device: Piezo-ICSI — During piezo-ICSI, a piezo-electric effect is generated through the conversion of electric energy to mechanical energy. This causes a smooth movement of the injection pipette, which allows for steady, controlled microinjection of a sperm with less psychical stress applied on the oocytes than by the conventional technique.
  Arms: Piezo-ICSI

SUMMARY:
Intracytoplasmic sperm injection (ICSI) has successfully been used to treat both severe male infertility and fertilization failure since its introduction in the early 1990´s. During the procedure a single sperm is injected into the cytoplasm of an oocyte to achieve fertilization. This technique is intrusive, has a relatively long learning curve and variable operator performance.

A new injection technique called piezo-ICSI has recently been introduced. During piezo-ICSI, a piezo-electric effect is generated through the conversion of electric energy to mechanical energy. This causes a smooth movement of the injection pipette, which allows for steady, controlled microinjections with less psychical stress applied on the oocytes than by the conventional technique.

A recent analysis, based on data from 9 different studies comparing conventional ICSI and piezo-ICSI (17500 cases), showed a benefit of piezo. Unfortunately, proper randomized trials are missing from this analysis. The proposed study is a randomized controlled study carried out at two private IVF clinics. Eligible participants are patients undergoing ICSI treatment, with a minimum of 6 oocytes. The participants will act as their own controls, with their oocytes randomly and equally divided between injection by the investigated and the conventional technique.

Whether piezo-ICSI is associated with improved success rates or reduction in adverse outcomes is at present unclear. Patients with fragile oocytes may benefit more from piezo-ICSI. In patients above 35 years, piezo-ICSI has been associated with a lower oocyte degeneration rate and an increased blastocyst rate. The aim of the study is to investigate whether the piezo-ICSI technique will result in more oocytes becoming normally fertilized compared to conventional ICSI. Another proposed benefit of piezo-ICSI lies in the standardization and simplification of the ICSI procedure. Making the injection procedure more independent of operator skill may result in a more robust and predictable laboratory output.

ELIGIBILITY:
Inclusion Criteria:

1. Patients receiving controlled ovarian stimulation with gonadotrophins needing ICSI for fertilizing oocytes.
2. Availability of at least six mature oocytes (MII) after oocyte pick-up.
3. Planned blastocyst culture.

Exclusion Criteria:

1. Intention to perform any form of preimplantation genetic testing
2. The use of IMSI or polarized light in the ICSI process
3. The use of assisted hatching prior to randomization.
4. Surgical sperm retrieval (SSR) patients.
5. Previous participation in this RCT
6. Concurrent participation in another investigation that can affect the primary outcome of this study.
7. Sperm sample with <0.1million/ml or motility of <2% after preparation.
8. Fertility preservation cycles.
9. If a day 2-4 transfer is planned
10. Use of vitrified oocytes.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 265 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Fertilization rate | Oocytes will be observed over a period of 26 hours after the intervention
  Number of normally fertilized oocytes per injected oocytes

SECONDARY OUTCOMES:
Percentage of degenerated oocytes | Oocytes will be observed over a period of 26 hours after the intervention
  Number of oocytes that have degenerated after the procedure
Percentage of 0 PN oocytes | Oocytes will be observed over a period of 26 hours after the intervention
  Number of oocytes not fertilized (0 PN) after the procedure.
Percentage of 1 PN oocytes. | Oocytes will be observed over a period of 26 hours after the intervention
  Number of oocytes fertilized with one pronuclei (1 PN) after the procedure.
Percentage of >2PN oocytes. | Oocytes will be observed over a period of 26 hours after the intervention
  Number of oocytes fertilized with more than 2 pronuclei (>2PN) after the procedure.
Differences in KID scores. | Embryos will be observed over a period of 6 days after the procedure
  Embryo development will be analysed using a mathematical models called KID (0-10 scale).
Differences in iDA scores. | Embryos will be observed over a period of 6 days after the procedure
  Embryo development will be analyzed using a artificial intelligence model, called iDA (0-10 scale).
Blastocyst rate (number of grade 3 or higher). | Embryos will be observed over a period of 6 days after the procedure
  Number of blastocysts with a morphological score of grade 3 or higher.
Percentage of cryopreserved blastocysts on day 5 and 6. | Embryos will be observed over a period of 6 days after the procedure
  Number of blastocysts cryopreserved on day 5 and day 6.
8. Utilization rate (Number of transferred and cryopreserved blastocysts). Utilization rate | Embryos will be observed over a period of 6 days after the procedure
  Number of transferred and cryopreserved blastocysts

CONTACTS AND LOCATIONS:
Overall Officials: Scott Nelson, MD, PhD, Principal Investigator — University of Glasgow
Locations (2):
- United Kingdom (2):
  - Nurture Fertility (TFP), Nottingham
  - Oxford Fertility (TFP), Oxford

IPD SHARING:
Plan to Share IPD: No